CLINICAL TRIAL: NCT01092520
Title: Open Label Pilot Study of Gabapentin for the Treatment of Pruritus Caused by Burn Injuries in Children
Brief Title: Gabapentin for the Treatment of Pruritus Caused by Burn Injuries in Children
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Jason Hayes, Staff Anesthesiologist, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1000013007
Record Dates: First submitted 2010-03-23; First posted 2010-03-25 (Estimated); Last update posted 2013-08-20 (Estimated); Status verified 2013-08

CONDITIONS: Pruritus
Keywords: Gabapentin; Burn Injuries in Children; pruritus
MeSH Terms: conditions — Pruritus | interventions — Gabapentin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gabapentin (Experimental)
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Gabapentin — Day 1 - 5mg/kg/dose per os at bedtime then 5mg/kg/dose PO b.i.d x 1 day (Day 2) then on Day 3, 5mg/kg/dose PO t.i.d . x 19 days; after 7 days, if not at maximal effect may increase over 3 days to 10mg/kg/dose (Day 8: 5 mg/kg/dose q.am and midday, Day 9: 10mg/kg/dose b.i.d. + 5mg/kg/dose midday, Day 10: 10mg/kg/dose t.i.d.) Doses may be reduced if patient experiences intolerable side effects.

SUMMARY:
Children with healing burns often suffer from pruritus that may continue for many months. Pruritus can be very distressing to the child and can interfere with sleep, activities of daily living, and rehabilitation therapy. Additionally, constant scratching of skin grafts may result in damage that requires further surgery, thus putting the patient at additional risk and adding to health care costs. Although the size of the burn injury is a risk factor for pruritus, almost 50% of patients with small burn injuries reported moderate or severe pruritus.

DETAILED DESCRIPTION:
Gabapentin has been shown to be effective for the treatment of pruritus in adult patients with brachioradial pruritus, uraemic pruritus and pruritus of unknown origin. Although the specific mechanism is unknown, the end result is the downregulation of excitatory neurotransmitter release and decrease in neuronal hyperexcitability.

The primary objective of this study is evaluating the effectiveness of gabapentin in reducing the severity of pruritus in children with burn injuries.

ELIGIBILITY:
Inclusion Criteria:

1. Children with partial or deep thickness burn
2. Children receiving triple antihistamines for treatment of pruritus
3. Children with a pruritus score ≥ 2 (Appendix 1) despite triple antihistamine therapy
4. Children who are tolerating liquids by mouth or nasogastric tube

Exclusion Criteria

1. Children with a medical condition for which gabapentin is contraindicated including children who have demonstrated a hypersensitivity to gabapentin or any of the components of the formulation.
2. Children with seizure disorders
3. Children with a pre-existing behavioural or developmental disorder
4. Children with renal impairment
5. Children with severe burns requiring PICU admission

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2009-07; Primary Completion 2011-07 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Pruritus score | Daily until discharge
  4-point scale validated in children 6 to 18 years of age, with additional descriptors from a similar scale used in adults

SECONDARY OUTCOMES:
Quality of Life Score | Daily until discharge
  Measured by the Children's Dermatology Quality Index
Antihistamine use | Daily until discharge or cessation of antihistamines
Opioid Consumption | Daily until discharge or cessation of opioid intake

CONTACTS AND LOCATIONS:
Overall Officials: Jason Hayes, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada